CLINICAL TRIAL: NCT03714633
Title: Stockholm Preterm Interaction-Based Intervention
Acronym: SPIBI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Karolinska Institutet (Other); Region Stockholm (Other Government); Centrum för kompetensutveckling inom vård och omsorg, Stockholm University (funding) (Unknown); Clas Groschinskys Minnesfond, Sweden (funding) (Unknown); Queen Silvia Jubilee Fund for research on children and disability, Sweden (funding) (Unknown); Filénska fonden, Sweden (funding) (Unknown)
Responsible Party: Principal Investigator, Professor Mara Westling Allodi, Professor in Special Education, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TiSam
Record Dates: First submitted 2018-09-26; First posted 2018-10-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Extreme Prematurity
Keywords: cognitive development; motor development; parent-child interaction; parental mental health; strength-based intervention; prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor of the parent-child interaction using the emotional availability scales is blind to if the child belongs to the intervention Group or Control Group. Several outcomes are self assessment questionnaires, with no masking.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stockholm Preterm Interaction-Based Intervention (SPIBI) (Experimental): Home-based post-discharge intervention for extreme premature babies and their parents. The intervention consists of one hospital visit, nine home-visits and two telephone calls during the first year corrected age, specifically from one week before discharge to 12 months corrected age. The intervention is strengths-based working with the infant-parent interaction, supporting infant development and strengthening the parent in his/her role.
  Interventions: Behavioral: Stockholm Preterm Interaction-Based Intervention (SPIBI)
- Control (No Intervention): The participants of the Control Group receives treatment as usual, which consists of a regular follow-up program with neurodevelopmental assessment at term age, 3 months corrected age, 12 months corrected age, 24 months corrected age and 66 months corrected age. Compared to children not participating in the study, the control group will receive an extended follow-up program, with assessment and questionnaires at term age, 3 months corrected age, 12 months corrected age, 24 months corrected age and 36 months corrected age. Participants in the control group will be referred to specialized care when needed.

INTERVENTIONS:
Behavioral: Stockholm Preterm Interaction-Based Intervention (SPIBI) — Post-discharge intervention to extreme premature infants and their parents
  Arms: Stockholm Preterm Interaction-Based Intervention (SPIBI)

SUMMARY:
Extreme premature Children will at discharge from Karolinska Hospital and Södersjukhuset in Stockholm be asked to participate in a study, examining the effects of a home-visit based post-discharge program aiming at facilitating the interaction between infants and parents, improving the development of the children, and the parental mental health. The study is a randomized controlled Trial (RCT), hence 50% of the participants will be offered treatment as usual (TAU) with addition of an extended follow-up program. The interaction-based program consists of one initial visit at the hospital followed by nine home-visits and two telephone calls during the child's first year of life. The interventionists are skilled Healthcare professionals with several years of experience from caring for premature infants and their parents. All interventionists have successfully completed a one year further education program, delivered one day per week and containing theoretical lectures, practice with actual cases, supervision on the cases, visits to the different parts of the neonatal care chain and discussions with a representative from the premature family association Sweden.

DETAILED DESCRIPTION:
Detailed description of the intervention: the purpose of the initial visit at the neonatal unit or hospital ward where the child is still treated is to establish the foundation for the interventionist/family relationship and give the parent(-s) the opportunity to show the interventionist the environment where the infant has spent his/her first 3-5 months in life.

Home-visit 1-3 and two telephone calls are provided before the child is three months corrected age. The focus of these home visits is to observe child and parent at home and validate the child's strengths and competences as well as enhancing the parent-child interaction, building on strengths. The child's strengths and interests will be summarized in a logbook owned by the parents. During home-visit 4-8 the interventionist, step by step and always with great regard to the child's level of development, will support the parent in using the home-environment in a developmental supporting manner for the child, find suitable objects/toys at home for the child to examine with mouth, hands and body, confirm the child's abilities and give suggestions on how to stimulate the child's further development. The logbook will now also contain suggestions for supporting the next developmental step, which will be formulated by the interventionist together with the parent. The ninth and last home-visit will emphasize the child's progress during the past year, look through the family logbook and both summarize the past year and talk about the next developmental step for the future.

The intervention group receives the standard follow-up program just as the control group and will be referred to specialized care when needed. Compared to children not participating in the study, the study participants will receive an extended follow-up program, with assessment and questionnaires at term age, 3 months corrected age, 12 months corrected age, 24 months corrected age and 36 months corrected age. The research process and the study protocol have been published, see references below.

ELIGIBILITY:
Inclusion Criteria:

* extremely premature born babies
* close to discharge from their neonatal intensive care unit hospital stay at Stockholm county council (Stockholms Läns Landsting).

Exclusion Criteria:

* Children with parent/parents who do not communicate in Swedish or English.
* Patients not residing in Stockholm county.
* Acute surgery patients who will spend a lot of time at hospitals far from Stockholm

Ages: 32 Weeks to 45 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 130 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-01-03 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Parent-child interaction | 12 months corrected age.
  Emotional availability scales, EAS The scale has four parental dimensions; sensitivity, structure, non-intrusiveness, non-hostility and two child dimensions; child responsiveness and child involvement. Each subscale has a maximum score of 29 and a direct score of 1-7. Hypothesis of higher scores in intervention group.

SECONDARY OUTCOMES:
Child's general development | 24 months corrected age
  Bayley scales of infant and toddler development (third edition; Bayley-III), measuring cognition, language, and motor development. Composite scores are standardized to mean (SD) scores of 100 (15), based on age-matched normative data. Higher scores in intervention group
Child's executive function | 24 and 36 months corrected age
  Behaviour Rating of Executive Function Parental version BRIEF-P. All the 5 subscales will be used. Hypothesis of less executive problems in intervention group.
Child's motor development 1 | 3 months & 12 months corrected age
  Alberta Infant Motor Scale, AIMS. Range 0 - 58 points, with a hypothesis of higher scores for intervention group
Parental depression | Term age, 12, 24 and 36 months corrected age
  Hospital anxiety and depression scale, HADS. Range depression subscale 0-21, range anxiety subscale 0-21. Hypothesis of lower scores in the intervention-parental group.
Parental anxiety | Term age, 12, 24 and 36 months corrected age
  State/trait anxiety inventory, STAI. Maximum 80 points for the State-scale, and maximum 80 points for the trait-scale. Hypothesis of lower scores in the intervention-parental group
Parental self-efficacy | Term age, 12, 24 and 36 months corrected age
  parental self-efficacy scale, PSE. PSE has 24 items at term age and 12 and 24 months and 48 items int he form for older ages, all items rated in a 0-10 scale. Hypothesis of higher score for intervention group at 12,24 and 36 months.
Parental resilience | Term age, 12, 24 and 36 months corrected age
  Resilience scale, RES. RES is a 25-items scale with a 7-point Likert scale. Hypothesis of higher scores in the intervention group.

OTHER OUTCOMES:
Child's neurological development | 3 months, 12 months, 24 months corrected age, hypothesis of higher score for intervention group
  Hammersmith infant neurological examination, range 0-78 with a hypothesis of higher scores in intervention group.
Child's motor development 2 | Term age & 12 months corrected age, hypothesis of higher score for intervention group
  Peabody developmental motor scales, PDMS. Subscale Stationary: range 0-42, subscale Locomotion range 0-138, subscale Object Manipulation range 0-30, subscale Grasping range 0-44 and subscale Visual-Motor Integration range 0-113. Hypothesis of higher scores in intervention group.
Child's motor development 3 | 3 months corrected age
  General movement assessment, GMA, scale Normal-Absent Fidgety
Child's general development | 12 months, 24 months, 36 months corrected age, hypothesis that the parents of the intervention group scoring their children higher
  Ages and stages questionnaire, ASQ-R. All five subscales Communication, Gross Motor, Fine Motor, Problem Solving, Personal-Social will be used, with a range from 0-300 all together. Hypothesis of higher scores in intervention group.
Child's strengths and difficulties | 24 and 36 months corrected age, hypothesis of less difficulties and more strengths scored by parents in the intervention group
  Strengths and difficulties questionnaire SDQ. 25 items on a 3-point scale, 5 questions of prosocial behaviour and 20 questions about various difficulties. Hypothesis of higher scores in the intervention group for prosocial behaviour and lower scores in the intervention group of the problematic subscales.
Child's autistic symptoms | 24 months corrected age
  Modified checklist for autism in toddlers M-CHAT. Range 0-20 points, hypothesis of lower scores in intervention group.
Infant temperament | 12 months corrected age
  Infant behavior questionnaire, IBQ-R. 37 items on a 7 point scale. Hypothesis of less problematic behaviour in intervention group, i.e. higher scores on subscales Smiling and Laughter and soothability; and lower scores on the subscales Fear and Distress to Limitations.
Parental satisfaction with the intervention | 12 months corrected age
  Client satisfaction questionnaire, CSQ-8 & semi-structured interview. CSQ-8 has 8 items, and a range of 8-48 points.
Pre-school educators' view of the child's engagement in preschool | 24 and 36 months corrected age
  Child Engagement Questionnaire (CEQ) Swedish version has 29 items rated on a 4 point scale and the summary score may range from 29 to 116 with higher scores indicating more positive engagement
Pre-school educators' view of the child's interaction in preschool | 24 and 36 months corrected age
  Swedish questionnaire Ert Barn Vårt Samspel, has 36 items rated on a 5 points scale and the summary score may range from 36 to 180 with higher scores indicating more interactive behavior
Pre-school educators' view of the child's playtime in preschool | 24 and 36 months corrected age
  Play time / Social Time Teacher Impression Scale. 16 items 1-5 Likert scale (min 16- max 80) higher scores indicating more social skills and play behavior
Pre-school educators' view of the child in preschool | 24 or 36 months corrected age, depending on when the child has entered preschool
  Semi-structured preschool teacher interview
Pre-school educators' view of the child's level of function in preschool | 24 and 36 months corrected age
  ICF-CY core sets. 12 items in Body functions (rated 0-9) and 22 items (rated 0-9) in Activities and Participation; higher scores indicate disability or developmental delay. 20 items covering Environmental factors (between +4 and +1 for facilitators; 0-9 for barriers) measure included to identify possible disability and environmental moderators.
Parent-child interaction long-term | 24 months corrected age
  Emotional availability scales, EAS The scale has four parental dimensions; sensitivity, structure, non-intrusiveness, non-hostility and two child dimensions; child responsiveness and child involvement. Each subscale has a maximum score of 29 and a direct score of 1-7. Hypothesis of higher scores in intervention group.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Ådén, MD PhD, Principal Investigator — Karolinska Institutet
Locations (5):
- Sweden (5):
  - Karolinska Hospital, Danderyds Sjukhus neonatalavdelning, Danderyd
  - Karolinska Hospital Huddinge, neontalavdelningen, Huddinge
  - Karolinska Hospital, Solna
  - Stockholm University, Stockholm
  - Södersjukhusets neonatalavdelning, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Verkerk G, Jeukens-Visser M, Houtzager B, Koldewijn K, van Wassenaer A, Nollet F, Kok J. The infant behavioral assessment and intervention program in very low birth weight infants; outcome on executive functioning, behaviour and cognition at preschool age. Early Hum Dev. 2012 Aug;88(8):699-705. doi: 10.1016/j.earlhumdev.2012.02.004. Epub 2012 Mar 10. PMID 22406323
- [Background] Koldewijn K, Wolf MJ, van Wassenaer A, Meijssen D, van Sonderen L, van Baar A, Beelen A, Nollet F, Kok J. The Infant Behavioral Assessment and Intervention Program for very low birth weight infants at 6 months corrected age. J Pediatr. 2009 Jan;154(1):33-38.e2. doi: 10.1016/j.jpeds.2008.07.039. Epub 2008 Sep 10. PMID 18783797
- [Background] Koldewijn K, van Wassenaer A, Wolf MJ, Meijssen D, Houtzager B, Beelen A, Kok J, Nollet F. A neurobehavioral intervention and assessment program in very low birth weight infants: outcome at 24 months. J Pediatr. 2010 Mar;156(3):359-65. doi: 10.1016/j.jpeds.2009.09.009. Epub 2009 Nov 2. PMID 19880139
- [Background] Meijssen DE, Wolf MJ, Koldewijn K, van Wassenaer AG, Kok JH, van Baar AL. Parenting stress in mothers after very preterm birth and the effect of the Infant Behavioural Assessment and Intervention Program. Child Care Health Dev. 2011 Mar;37(2):195-202. doi: 10.1111/j.1365-2214.2010.01119.x. PMID 20645992
- [Background] Spittle A, Orton J, Anderson PJ, Boyd R, Doyle LW. Early developmental intervention programmes provided post hospital discharge to prevent motor and cognitive impairment in preterm infants. Cochrane Database Syst Rev. 2015 Nov 24;2015(11):CD005495. doi: 10.1002/14651858.CD005495.pub4. PMID 26597166
- [Background] Baraldi E, Allodi MW, Lowing K, Smedler AC, Westrup B, Aden U. Stockholm preterm interaction-based intervention (SPIBI) - study protocol for an RCT of a 12-month parallel-group post-discharge program for extremely preterm infants and their parents. BMC Pediatr. 2020 Feb 1;20(1):49. doi: 10.1186/s12887-020-1934-4. PMID 32007087
- [Background] Baraldi, E., Westling Allodi, M., Löwing, K., Smedler, A.-C., Westrup, B., & Ådén, U. (2019). Clinical Protocol & Research Process of Stockholm Preterm Interaction-Based Intervention, SPIBI. Pediatric Research, 86(Suppl.), 54-55. https://doi.org/10.1038/s41390-019-0521-6
- [Result] Baraldi E, Allodi MW, Smedler AC, Westrup B, Lowing K, Aden U. Parents' Experiences of the First Year at Home with an Infant Born Extremely Preterm with and without Post-Discharge Intervention: Ambivalence, Loneliness, and Relationship Impact. Int J Environ Res Public Health. 2020 Dec 13;17(24):9326. doi: 10.3390/ijerph17249326. PMID 33322234
- See also: Link to project information — https://www.su.se/english/research/research-projects/stockholm-preterm-interaction-based-intervention-spibi?open-collapse-boxes=research-project-publications,research-project-members,research-project-description